CLINICAL TRIAL: NCT03059602
Title: Characterizing the Biopsychosocial Impact on Caregivers in Patients Undergoing Joint Replacement and Cervical/Thoracic/Lumbar Spine Surgery: A Pilot Study
Brief Title: Biopsychosocial Impact on Caregivers in Patients Undergoing Joint and Spine Surgery
Status: Completed | Type: Observational
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Responsible Party: Sponsor
Other Study IDs: 500115
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Knee group: Caregivers who will be the primary source of assistance (medical, rehabilitative, daily living, etc) after surgery for patients undergoing total knee arthroplasty.
  Interventions: Other: No specific treatment based intervention-health measurement instrument
- Hip group: Caregivers who will be the primary source of assistance (medical, rehabilitative, daily living, etc) after surgery for patients undergoing total hip arthroplasty.
  Interventions: Other: No specific treatment based intervention-health measurement instrument
- Spine group: Caregivers who will be the primary source of assistance (medical, rehabilitative, daily living, etc) after surgery for patients undergoing Cervical/Thoracic Lumbar Spine Surgery (Discectomy, Foraminotomy, Laminectomy, Fusion, Nerve Root Decompression)
  Interventions: Other: No specific treatment based intervention-health measurement instrument

INTERVENTIONS:
Other: No specific treatment based intervention-health measurement instrument — Caregivers will receive a series of standard health measurement tools/survey from NIH's Patient Reported Outcome Measurement Information System (PROMIS)

SUMMARY:
The purpose of this study is to describe the biopsychosocial impact of caregivers in patients undergoing total knee arthroplasty, total hip arthroplasty, and cervical/thoracic/lumbar spine surgery.Defining such impacts may offer opportunities to enhance caregiver capability to provide care following surgery on a loved one.

DETAILED DESCRIPTION:
This is a pilot feasibility study with the goal of enrolling 50 caregivers in each surgical subgroup, with a total of 150 subjects. Caregivers for patients undergoing the above surgeries will be administered Patient Reported Outcome Measurement Information System (PROMIS) measures preoperatively, 7 days postoperatively, 14 days postoperatively, and 1 month postoperatively. PROMIS item banks will include Global Health, Anxiety, Fatigue, Depression, Self Efficacy, Social Satisfaction, and Sleep Disturbance. If the caregiver reports the presence of persistent pain, Pain Interference and Physical Function will be administered.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Are the primary person helping in the recovery of a patient undergoing one of the following surgeries below with in the first 30 days after surgery Total knee arthroplasty Total hip arthroplasty Cervical/Thoracic/Lumbar spine surgery
* Able to understand English and can verbalize their pain level

Exclusion Criteria:

* Younger than 18 years old
* Refuse participation
* Cannot understand English
* Has cognitive deficiencies (subject unable to provide consent for the study, subject unable to complete initial post consent measures)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregivers of male and female military health care beneficiaries age 18 years and older presenting for total knee arthroplasty, total hip arthroplasty, and Cervical/Thoracic/Lumbar spine surgery. Caregivers are defined as individuals who will be the primary source of assistance (medical, rehabilitative, daily living, etc) within the first 30 days after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Natural history of biopsychosocial impact of Caregivers | 1 month
  To describe the natural history of the biopsychosocial impact of Caregivers for patients undergoing total knee arthroplasty, total hip arthroplasty, and cervical/thoracic/lumbar spinal surgery.

SECONDARY OUTCOMES:
Change of biopsychosocial measures over time | 1 month
  To assess the biopsychosocial measure over time from the following time points: Preoperative, 7 days, 14 days postoperatively, and 1 month postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No